CLINICAL TRIAL: NCT03960190
Title: Clinical Investigation to Assess the Performance of the Eureka Electric Breast Pump in Mothers Breastfeeding Their Healthy Term Infant
Acronym: EUREKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Consumer Lifestyle (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HW-MCC-Eureka-2019-10559
Record Dates: First submitted 2019-05-15; First posted 2019-05-22 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Breast Pumping
MeSH Terms: conditions — Breast Milk Expression

STUDY DESIGN:
Intervention Model Description: The Investigational Device used for this study, is an electric breast pump, intended to express and collect milk from the breast of a lactating woman. Both the 1K and 2K expression kit will be tested in single and double pumping regime.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1K expression kit (Experimental): Subjects will be using the breastpump with the with 1K expression kit.
  Interventions: Device: Using Eureka Breast Pump with Expression Kit
- 2K expression kit (Experimental): Subjects will be using the breastpump with the with 2K expression kit.
  Interventions: Device: Using Eureka Breast Pump with Expression Kit

INTERVENTIONS:
Device: Using Eureka Breast Pump with Expression Kit — Each subject will undergo two expression sessions for single and double electric pumping in randomized order to reduce the variation.

SUMMARY:
Babies are the best in class in order to get human milk out of a lactating breast. With this in mind, Philips has developed the a new electric breast pump, attempting to mimic the babies sucking behavior. The new electric breast pump includes a new vacuum profile and 2 new expression kits.

DETAILED DESCRIPTION:
Breast pumps currently on the market function by applying vacuum directly to the breast. The effect of a build-up of pressure within the breast due to the accumulation of milk, combined with the external negative pressure introduced by the breast pump, results in the expression of milk. However, in order to express sufficient amounts of milk it is important to stimulate the Milk Ejection Reflex (MER). The MER, also called letdown, draught ejection, expulsion or pumping reflex, is described as a response of the mammary gland to oxytocin. When the nipple is stimulated, the mother's posterior pituitary gland releases oxytocin into the bloodstream. Upon reaching the breast tissue, oxytocin provokes contraction of cells within the structure of the breast causing milk flow. Without the MER successful breastfeeding or breast milk expression cannot happen. In order to stimulate the MER, Philips has developed 2 new expression kits to better mimic the suckling pattern of an infant.

ELIGIBILITY:
Inclusion Criteria:

* Have an age between 18 and 50 years
* Have delivered a healthy, term singleton infant (with birth weight above 2.5kg and at least 37 weeks gestation)
* Have a baby with an age between 1 and 4 months
* Exclusively breastfeeding at the time of the study
* Have signed the Informed Consent form

Exclusion Criteria:

* Pregnant at the time of the study
* Suffer from known side effects (sore nipples, nipple trauma, bruising, engorgement, clogged mammary ducts, lactostasis, mastitis) at the time of the study
* Suffer from syndrome of Raynaud
* When providing complementary foods to their baby at the time of the study
* When providing donor milk and/or formula milk to their baby at the time of the study
* When having their period at the time of the study
* When taking oral anticonception at the time of the study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Breast feeding women
Enrollment: 40 (Actual)
Dates: Start 2019-05-17 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2019-10-22 (Actual)

PRIMARY OUTCOMES:
Evaluating the performance via percentage of the end milk weight that is expressed during the first 5 minutes after pump start of the Eureka electric breast pump and 1K and 2K expression kits. | 3 months
  The data of the expression sessions will be averaged within each of the single and double pumping regimes.

SECONDARY OUTCOMES:
Evaluating the performance weight of expressed milk at 1-minute intervals of the Eureka electric breast pump and 1K and 2K expression kits. | 3 months
  The data of the expression sessions will be averaged within each of the single and double pumping regimes.
Evaluating the performance via total expression time in minutes of the Eureka electric breast pump and 1K and 2K expression kits. | 3 months
  The data of the expression sessions will be averaged within each of the single and double pumping regimes.
Evaluating the performance of time to first milk ejection reflex (MER) pump in seconds of the Eureka electric breast pump and 1K and 2K expression kits. | 3 months
  The data of the expression sessions will be averaged within each of the single and double pumping regimes.
Evaluating the performance via weight (grams) of expressed milk after full expression session of the Eureka electric breast pump and 1K and 2K expression kits. | 3 months
  The data of the expression sessions will be averaged within each of the single and double pumping regimes.

CONTACTS AND LOCATIONS:
Locations (1):
- Philips Innovation Site Eindhoven, Eindhoven, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Health Organzation: http://www.who.int/topics/breastfeeding/en/.
- [Background] Victora CG, Bahl R, Barros AJ, Franca GV, Horton S, Krasevec J, Murch S, Sankar MJ, Walker N, Rollins NC; Lancet Breastfeeding Series Group. Breastfeeding in the 21st century: epidemiology, mechanisms, and lifelong effect. Lancet. 2016 Jan 30;387(10017):475-90. doi: 10.1016/S0140-6736(15)01024-7. PMID 26869575
- [Background] Zoppou C, Barry SI, Mercer GN. Dynamics of human milk extraction: a comparative study of breast feeding and breast pumping. Bull Math Biol. 1997 Sep;59(5):953-73. doi: 10.1007/BF02460001. PMID 9281906
- [Background] Riordan J, Gill-Hopple K, Angeron J. Indicators of effective breastfeeding and estimates of breast milk intake. J Hum Lact. 2005 Nov;21(4):406-12. doi: 10.1177/0890334405281032. PMID 16280556